CLINICAL TRIAL: NCT04406246
Title: Prevention of Coronavirus Disease (COVID-19) Outbreaks by Prophylactic Treatment With Nitazoxanide
Brief Title: Prevention of Coronavirus Disease (COVID-19) Outbreaks With Nitazoxanide
Status: Completed | Phase: Phase 4 | Type: Interventional
Sponsor: Materno-Perinatal Hospital of the State of Mexico (Other)
Collaborators: Laboratorios Liomont (Industry)
Responsible Party: Principal Investigator, Hugo Mendieta Zeron, Chief of the Research Department, Materno-Perinatal Hospital of the State of Mexico
Allocation: Not Applicable | Model: Single Group | Masking: None | Purpose: Treatment
Other Study IDs: 2020-04-682
Record Dates: First submitted 2020-05-24; First posted 2020-05-28 (Actual); Last update posted 2021-03-30 (Actual); Status verified 2021-03

CONDITIONS: Coronavirus Infection
Keywords: evolution; nitazoxanide
MeSH Terms: conditions — Coronavirus Infections | interventions — nitazoxanide; Tablets

STUDY DESIGN:
Intervention Model Description: In this cohort study, all health workers of the Maternal-Perinatal Hospital "Mónica Pretelini Sáenz", with symptoms of SARS-CoV-2 will be treated promptly with nitazoxanide.
Oversight: Data Monitoring Committee: Yes | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (1):
- Nitazoxanide early treatment (Experimental): Health workers with symptoms of COVID-19 not requiring hospitalization will receive an early treatment with nitazoxanide.
  Interventions: Drug: Nitazoxanide 500Mg Oral Tablet

INTERVENTIONS:
Drug: Nitazoxanide 500Mg Oral Tablet — Health workers affected by SARS-CoV-2 will receive the next doses of nitazoxanide: 500 mg every 6 hour for two days and then every 12 hours for four days.
  Other Names: Paramix

SUMMARY:
The new coronavirus outbreak has led to a public health emergency of international concern, putting all health organizations on high alert. As part of the hygienic measures, isolation and reinforcement cleaning strategies have been followed. It is known that special attention and efforts should be applied to protect or reduce transmission in susceptible populations, including the elderly or those with comorbidities.It has also been proposed a semaforization to classify patients with respiratory symptoms based on: Fever (38ºC or more), dry cough, headache, dyspnea, joint pain, muscle pain, sore throat, nose discharge, conjunctivitis, chest pain, diarrhea, anosmia, ageusia.

Nitazoxanide has shown to be effective against several viruses, of both types RNA and DNA, including other coronavirus that produced the Severe Acute Respiratory Syndrome (SARS) and the Middle East Respiratory Syndrome (MERS).

Facing the lack of options against COVID-19 outbreaks for example in health workers, nitazoxanide could contribute to decrease the contagious dissemination of SARS-CoV-2, thus reducing at the same time the Hospital saturation of patients positive to this virus.

DETAILED DESCRIPTION:
Coronaviruses (CoV) are positive-stranded single-stranded RNA viruses that infect a wide range of hosts. The new coronavirus outbreak has led to a public health emergency of international concern, putting all health organizations on high alert.

The accelerated spread pushed physicians to try a variety of treatments without an established sequence due to ignorance of the disease. As part of the hygienic measures, isolation and reinforcement cleaning strategies have been followed. With current epidemiological data, it is known that special attention and efforts should be applied to reduce the transmission in susceptible populations, including the elderly or those with comorbidities. On the other hand it has also been proposed a semaforization to classify the severity of COVID-19 cases.

Nitazoxanide, a drug with antibacterial and anti-protozoal effects, has also powerful antiviral effects through the phosphorylation of protein-kinase activated by double-stranded RNA, which leads to an increase in phosphorylated factor 2-alpha, an intracellular protein with antiviral effects. This drug has been effective in vitro against Severe Acute Respiratory Syndrome (SARS) and Middle East Respiratory Syndrome by Coronavirus (MERS), both produced by other coronavirus.

Currently all the efforts in the world have been focused on the treatment of COVID-19 since there is pneumonia, the patient being in hospitalization and even in intensive care units. Probably, focusing on these late stages has distracted the attention of the initial stage, this means early treatment to prevent the evolution to critical clinical conditions.

It is hypothesized that the use of nitazoxanide at an early stage of COVID-19 could decrease the contagious outbreaks of this virus in health workers, and at the same time will reduce the community dissemination and evolution of cases requiring intensive care units.

ELIGIBILITY:
Inclusion Criteria:

* COVID-19 positive patients by clinical criteria.

Exclusion Criteria:

* Patients who have inherent contraindications to nitazoxanide.
* Patients with inflammatory bowel disease.

Ages: 18 Years to 80 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 150 (Actual)
Dates: Start 2020-05-21 (Actual); Primary Completion 2020-12-31 (Actual); Study Completion 2020-12-31 (Actual)

PRIMARY OUTCOMES:
Health workers that require hospitalization | Two weeks since the begining of symptoms
  The percentage of health workers that require hospitalization after beginning an early treatment with nitazoxanide in case of referring symptoms of COVID-19.

CONTACTS AND LOCATIONS:
Overall Officials: José Meneses Calderón, MD., Principal Investigator — Research Unit
Locations (1):
- Materno-Perinatal Hospital "Mónica Pretelini", Toluca, Mexico

IPD SHARING:
Plan to Share IPD: Undecided
The Data will be available upon request after a publication is reached.

REFERENCES:
- [Background] Dhama K, Sharun K, Tiwari R, Dadar M, Malik YS, Singh KP, Chaicumpa W. COVID-19, an emerging coronavirus infection: advances and prospects in designing and developing vaccines, immunotherapeutics, and therapeutics. Hum Vaccin Immunother. 2020 Jun 2;16(6):1232-1238. doi: 10.1080/21645515.2020.1735227. Epub 2020 Mar 18. PMID 32186952
- [Background] Mifsud EJ, Tilmanis D, Oh DY, Ming-Kay Tai C, Rossignol JF, Hurt AC. Prophylaxis of ferrets with nitazoxanide and oseltamivir combinations is more effective at reducing the impact of influenza a virus infection compared to oseltamivir monotherapy. Antiviral Res. 2020 Apr;176:104751. doi: 10.1016/j.antiviral.2020.104751. Epub 2020 Feb 20. PMID 32088248
- [Background] Rossignol JF. Nitazoxanide, a new drug candidate for the treatment of Middle East respiratory syndrome coronavirus. J Infect Public Health. 2016 May-Jun;9(3):227-30. doi: 10.1016/j.jiph.2016.04.001. Epub 2016 Apr 16. PMID 27095301
- [Background] Rossignol JF. Nitazoxanide: a first-in-class broad-spectrum antiviral agent. Antiviral Res. 2014 Oct;110:94-103. doi: 10.1016/j.antiviral.2014.07.014. Epub 2014 Aug 7. PMID 25108173